CLINICAL TRIAL: NCT04004611
Title: A Multicenter, Open-Label PK Study of Mirikizumab in Pediatric Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Mirikizumab (LY3074828) in Children and Teenagers With Ulcerative Colitis (UC)
Acronym: SHINE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17410; I6T-MC-AMBU (Other: Eli Lilly and Company); 2019-001298-96 (EudraCT Number)
Record Dates: First submitted 2019-06-29; First posted 2019-07-02 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Ulcerative Colitis
Keywords: Interleukin-23 (IL-23) antibody; IL-23p19; Pediatric
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Open Label (OL) Induction Period: 5 milligram per kilogram (mg/kg) Miri intravenous (IV) (Experimental): Participants (≤40 kg weight) received 5 mg/kg mirikizumab given as an IV infusion every 4 weeks (Q4W) on weeks 0, 4, 8 for 12 weeks.
  Interventions: Drug: Mirikizumab
- Open Label Induction Period: 10 mg/kg Miri IV (Experimental): Participants (≤40 kg weight) received 10 mg/kg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks.
  Interventions: Drug: Mirikizumab
- Open Label Induction Period: 300 mg Miri IV (Experimental): Participants (>40 kg weight) received 300 mg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks.
  Interventions: Drug: Mirikizumab
- Open Label Maintenance Period: 50 mg Miri subcutaneous (SC) (Experimental): Participants (≤20 kg weight) who were responders to mirikizumab at week 12 in induction received 50 mg subcutaneously (SC) Q4W from week 12 through week 48 or until loss of response was confirmed.
  Interventions: Drug: Mirikizumab
- Open Label Maintenance Period: 100 mg Miri SC (Experimental): Participants (>20 to ≤40 kg weight) who were responders to mirikizumab at week 12 in induction received 100 mg SC Q4W from week 12 through week 48 or until loss of response was confirmed.
  Interventions: Drug: Mirikizumab
- Open Label Maintenance Period: 200 mg Miri SC (Experimental): Participants (>40 kg weight) who were responders to mirikizumab at week 12 in induction received 200 mg SC Q4W from week 12 through week 48 or until loss of response was confirmed.
  Interventions: Drug: Mirikizumab
- Open Label Maintenance Period: Non-Responders: 10 mg/kg Miri IV/ 50 mg Miri SC (Experimental): Participants (≤40 kg) who were non responders to miri at Week 12 in induction received 10 mg SC Q4W for 12 weeks or discontinued after repeat induction, and then received 50 mg miri (≤20 kg weight) SC Q4W through week 48 or until loss of response was confirmed.
  Interventions: Drug: Mirikizumab
- Open Label Maintenance Period: Non-Responders: 10 mg/kg Miri IV/100 mg Miri SC (Experimental): Participants (≤40 kg) who were non responders to miri at week 12 in induction received 10 mg SC Q4W for 12 weeks or discontinued after repeat induction, and then received 100 mg miri (>20 to ≤40 kg weight) SC Q4W through week 48 or until loss of response was confirmed.
  Interventions: Drug: Mirikizumab
- Open Label Maintenance Period: Non-Responders: 300 mg Miri IV /200 mg Miri SC (Experimental): Participants (>40 kg) who were non responders to miri at week 12 in induction received 300 mg SC Q4W for 12 weeks or discontinued after repeat induction, then received 200 mg miri SC Q4W through week 48 or until loss of response was confirmed.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered IV and SC
  Other Names: LY3074828

SUMMARY:
This study was designed to evaluate how the body processes and removes mirikizumab. The study also evaluated safety and disease response in pediatric participants with UC taking mirikizumab. The study lasted about 52 weeks and included up to 18 visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants weighing >10 kg
* Participants must have a diagnosis of ulcerative colitis for at least 3 months before the planned start date for the study medications
* Participants must have moderately to severely active UC as defined by a Modified Mayo Score (MMS) within 14 days before the first dose of study treatment
* Participants must have evidence of UC extending proximal to the rectum
* Participants must have demonstrated an inadequate response to, a loss of response to, or an intolerance to corticosteroids, immunomodulators, Janus kinase inhibitor (JAK-inhibitor) or to biologic therapies for UC

Exclusion Criteria:

* Participants must not have a current diagnosis of Crohn's disease, inflammatory bowel disease-unclassified (indeterminate colitis), ulcerative proctitis, or primary sclerosing cholangitis
* Participants must not have had surgery to remove part of their colon
* Participants must not have current evidence of toxic megacolon
* Participants must not have received any of the following for treatment of UC: cyclosporine or thalidomide within 30 days of screening; corticosteroid enemas, corticosteroid suppositories, or topical treatment with 5-aminosalicyclic acid within 1 week of screening endoscopy
* Participants must not have had an inadequate response to Interleukin-12 p40 subunit antibody (anti-IL12p40) (e.g. ustekinumab) or had prior exposure to anti-IL-23p19 antibodies (e.g. risankizumab, brazikumab, guselkumab or tildrakizumab)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (22):
  - Childrens Hospital of Orange County, Orange, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Children's Hospital of Colorado, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Emory University, Atlanta, Georgia
  - Children's Center for Digestive Health Care, LLC, Atlanta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Riley Hospital for Children, Carmel, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - MGH for Children - Waltham, Waltham, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Goryeb Children's Hospital / Atlantic Health System, Morristown, New Jersey
  - Icahn Sch of Med at Mt. Sinai, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - The Abbigail Wexner Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Cook Children's Hospital, Fort Worth, Texas
  - Texas Childrens Hospital, Houston, Texas
  - Pediatrics Specialists of Virginia, Fairfax, Virginia
  - Children's Hospital of The King's Daughters Inc, Norfolk, Virginia
  - Seattle Children's Hospital Research Foundation, Seattle, Washington
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto, Ontario
- Israel (3):
  - Rambam Medical Center, Haifa
  - The Juliet Keidan Institute of Paediatric Gastroenterology and Nutrition; Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
- Japan (7):
  - Kurume University Hospital, Kurume, Fukuoka
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Saitama Children's Medical Center, Saitama-shi, Saitama
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical and Dental University Hospital, Bunkyō, Tokyo
  - National Center For Child Health And Development, Setagaya-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
- South Korea (2):
  - Kyungpook National University Medical Center Chilgok Hospital, Daegu
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kaplan JL, Bousvaros A, Turner D, Dubinsky M, Larkin A, Johns J, Otani Y, Crandall W, Komocsar WJ, Hyams JS. Efficacy and safety of mirikizumab in paediatric participants with moderately-to-severely active ulcerative colitis (SHINE-1): a multicentre, open-label, non-randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2026 Feb;11(2):100-109. doi: 10.1016/S2468-1253(25)00196-7. Epub 2025 Nov 19. PMID 41270771
- See also: A Study of Mirikizumab (LY3074828) in Children and Teenagers With Ulcerative Colitis (UC) — https://trials.lillytrialguide.com/en-US/trial/2c0yudZdAogZJ3JBUHvV8U

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Mirikizumab (Miri) dose groups to which pediatric participants are assigned at week (wk) 0 (for induction period) and at wk 12 (for maintenance period) are dependent on participant' s weight and their clinical response status at wk 12 for maintenance period. All participants who achieved a modified Mayo score (MMS) clinical response at wk 12 or wk 24 [non-responders (NR) at wk 12 who received extended intravenous (IV) induction dosing for 12 more wks] were eligible for the maintenance period.
Groups:
- Open Label (OL) Induction Period: 5 Milligram Per Kilogram (mg/kg) Miri IV: Participants (≤40 kg weight) received 5 mg/kg mirikizumab given as an IV infusion every 4 weeks (Q4W) on weeks 0, 4, 8 for 12 weeks.
- OL Induction Period: 10 mg/kg Miri IV: Participants (≤40 kg weight) received 10 mg/kg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks.
- OL Induction Period: 300 mg Miri IV: Participants (>40 kg weight) received 300 mg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks.
- OL Maintenance Period: 50 mg Miri Subcutaneous (SC): Participants (≤20 kg weight) who were responders to mirikizumab at week 12 in induction received 50 mg SC Q4W from week 12 through week 48 or until loss of response was confirmed.
- OL Maintenance Period: 100 mg Miri SC: Participants (>20 to ≤40 kg weight) who were responders to mirikizumab at week 12 in induction received 100 mg SC Q4W from week 12 through week 48 or until loss of response was confirmed.
- OL Maintenance Period: 200 mg Miri SC: Participants (>40 kg weight) who were responders to mirikizumab at week 12 in induction received 200 mg SC Q4W from week 12 through week 48 or until loss of response was confirmed.
- OL Maintenance Period: NR: 10 mg/kg Miri IV/50 mg Miri SC: Participants (≤40 kg) who were non responders to miri at week 12 in induction received 10 mg SC Q4W for 12 weeks or discontinued after repeat induction, and then received 50 mg miri (≤20 kg weight) SC Q4W through week 48 or until loss of response was confirmed.
- OL Maintenance Period: NR: 10 mg/kg Miri IV/100 mg Miri SC: Participants (≤40 kg) who were non responders to miri at week 12 in induction received 10 mg SC Q4W for 12 weeks or discontinued after repeat induction, and then received 100 mg miri (>20 to ≤40 kg weight) SC Q4W through week 48 or until loss of response was confirmed.
- OL Maintenance Period: NR: 300 mg Miri IV /200 mg Miri SC: Participants (>40 kg) who were non responders to miri at week 12 in induction received 300 mg SC Q4W for 12 weeks or discontinued after repeat induction, then received 200 mg miri SC Q4W through week 48 or until loss of response was confirmed.
Period: OL Induction Period (Wk 0-12)
Arm/Group | Open Label (OL) Induction Period: 5 Milligram Per Kilogram (mg/kg) Miri IV | OL Induction Period: 10 mg/kg Miri IV | OL Induction Period: 300 mg Miri IV | OL Maintenance Period: 50 mg Miri Subcutaneous (SC) | OL Maintenance Period: 100 mg Miri SC | OL Maintenance Period: 200 mg Miri SC | OL Maintenance Period: NR: 10 mg/kg Miri IV/50 mg Miri SC | OL Maintenance Period: NR: 10 mg/kg Miri IV/100 mg Miri SC | OL Maintenance Period: NR: 300 mg Miri IV /200 mg Miri SC
Started | 10 | 5 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 10 | 5 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: OL Maintenance Period (Wk 12-52)
Arm/Group | Open Label (OL) Induction Period: 5 Milligram Per Kilogram (mg/kg) Miri IV | OL Induction Period: 10 mg/kg Miri IV | OL Induction Period: 300 mg Miri IV | OL Maintenance Period: 50 mg Miri Subcutaneous (SC) | OL Maintenance Period: 100 mg Miri SC | OL Maintenance Period: 200 mg Miri SC | OL Maintenance Period: NR: 10 mg/kg Miri IV/50 mg Miri SC | OL Maintenance Period: NR: 10 mg/kg Miri IV/100 mg Miri SC | OL Maintenance Period: NR: 300 mg Miri IV /200 mg Miri SC
Started | 0 (Participants were assigned to this arm only during open label induction period.) | 0 (Participants were assigned to this arm only during open label induction period.) | 0 (Participants were assigned to this arm only during open label induction period.) | 1 (Included only participants who entered open label maintenance period.) | 8 (Included only participants who entered open label maintenance period.) | 9 (Included only participants who entered open label maintenance period.) | 1 (Included only participants who entered open label maintenance period.) | 1 (Included only participants who entered open label maintenance period.) | 6 (Included only participants who entered open label maintenance period.)
Completed | 0 | 0 | 0 | 1 | 7 | 8 | 0 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Not completed — Withdrawal by Parent or Guardian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: OL Induction and Maintenance Period
Arm/Group | Open Label (OL) Induction Period: 5 Milligram Per Kilogram (mg/kg) Miri IV | OL Induction Period: 10 mg/kg Miri IV | OL Induction Period: 300 mg Miri IV | OL Maintenance Period: 50 mg Miri Subcutaneous (SC) | OL Maintenance Period: 100 mg Miri SC | OL Maintenance Period: 200 mg Miri SC | OL Maintenance Period: NR: 10 mg/kg Miri IV/50 mg Miri SC | OL Maintenance Period: NR: 10 mg/kg Miri IV/100 mg Miri SC | OL Maintenance Period: NR: 300 mg Miri IV /200 mg Miri SC
Started | 10 (Included only participants who entered open label induction and maintenance period.) | 5 (Included only participants who entered open label induction and maintenance period.) | 11 (Included only participants who entered open label induction and maintenance period.) | 0 (Participants were assigned to this arm only during open label maintenance period.) | 0 (Participants were assigned to this arm only during open label maintenance period.) | 0 (Participants were assigned to this arm only during open label maintenance period.) | 0 (Participants were assigned to this arm only during open label maintenance period.) | 0 (Participants were assigned to this arm only during open label maintenance period.) | 0 (Participants were assigned to this arm only during open label maintenance period.)
Completed | 9 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent or Guardian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- OL Induction Period: 5 mg/kg Miri IV: Participants (≤40 kg weight) received 5 mg/kg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | OL Induction Period: 5 mg/kg Miri IV | OL Induction Period: 10 mg/kg Miri IV | OL Induction Period: 300 mg Miri IV | Total
Number analyzed (Participants) | 10 | 5 | 11 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (4.22) | 11.6 (1.14) | 14.0 (1.26) | 11.80 (3.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 6 | 15
  Male | 4 | 2 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 2 | 3 | 8 | 13
  Unknown or Not Reported | 5 | 2 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 3 | 9 | 17
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Israel | 0 | 0 | 1 | 1
  Japan | 1 | 2 | 1 | 4
  South Korea | 4 | 0 | 0 | 4
  United States | 5 | 3 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Clearance of Mirikizumab
Description: Clearance of mirikizumab was evaluated. The PK of mirikizumab is characterized at interim analysis points using mixed-effect (population PK) modelling approaches using the available induction and maintenance mirikizumab concentration data.
Time Frame: Predose on week 4, 8, 12,16, 24, 36, 52 and post dose on week 0 and 8
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour per kilogram (L/hr/kg)
Groups:
- Mirikizumab: Participants weighing >40 kg received a mirikizumab induction dose of 300 mg via IV infusion and participants weighing ≤40 kg received induction doses of 5 or 10 mg/kg via IV infusion at weeks 0, 4, and 8 for 12 weeks.
Arm/Group | Mirikizumab
Number analyzed (Participants) | 26
Liters per hour per kilogram (L/hr/kg) | 0.000190 (59.74)

2. Secondary Outcome: Percentage of Participants in Clinical Remission
Description: Clinical remission at week 52 is defined as achieving a 9-point modified Mayo score (MMS) for rectal bleeding (RB) = 0, stool frequency (SF) = 0 or 1 and endoscopy (ES) = 0 or 1 (excluding friability). The MMS is a composite score of ulcerative colitis disease activity calculated as the sum of three subscores: SF subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal); RB subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed); ES subscore, based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding,ulceration.
Time Frame: Week 52
Population: Modified Intention-to-treat population (mITT): All randomized participants who received at least one dose of study drug and who had the clinical remission measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maintenance Period: 50 mg Miri SC Q4W: Participants (≤20 kg weight) who were responders to mirikizumab at week 12 in induction received 50 mg subcutaneously (SC) Q4W from week 12 through week 48 or until loss of response was confirmed.
- Maintenance Period: 100 mg Miri SC Q4W: Participants (>20 to ≤40 kg weight) who were responders to mirikizumab at week 12 in induction received 100 mg SC Q4W from week 12 through week 48 or until loss of response was confirmed.
- Maintenance Period: 200 mg Miri SC Q4W: Participants (>40 kg weight) who were responders to mirikizumab at week 12 in induction received 200 mg SC Q4W from week 12 through week 48 or until loss of response was confirmed.
- Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC: Participants (≤40 kg) who were non responders to miri at week 12 in induction received 10 mg SC Q4W for 12 weeks or discontinued after repeat induction, and then received 50 mg miri (≤20 kg weight) SC Q4W through week 48 or until loss of response was confirmed.
- Maintenance Period: 10 mg/kg Miri IV/100 mg Miri SC: Participants (≤40 kg) who were non responders to miri at week 12 in induction received 10 mg SC Q4W for 12 weeks or discontinued after repeat induction, and then received 100 mg miri (>20 to ≤40 kg weight) SC Q4W through week 48 or until loss of response was confirmed.
- Maintenance Period: 300 mg Miri IV/200 mg Miri SC: Participants (>40 kg) who were non responders to miri at week 12 in induction received 300 mg SC Q4W for 12 weeks or discontinued after repeat induction, then received 200 mg miri SC Q4W through week 48 or until loss of response was confirmed.
Arm/Group | Maintenance Period: 50 mg Miri SC Q4W | Maintenance Period: 100 mg Miri SC Q4W | Maintenance Period: 200 mg Miri SC Q4W | Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC | Maintenance Period: 10 mg/kg Miri IV/100 mg Miri SC | Maintenance Period: 300 mg Miri IV/200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
percentage of participants | 0.0 [0.0 to 79.3] | 62.5 [30.6 to 86.3] | 55.6 [26.7 to 81.1] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 39.0]

3. Secondary Outcome: Percentage of Participants in Clinical Response
Description: Clinical response at week 52 is defined as a decrease in the 9-point modified Mayo score (MMS) [rectal bleeding, stool frequency and the endoscopic findings] inclusive of ≥2 points and ≥30% from baseline with either a decrease of rectal bleeding subscore of ≥1 or rectal bleeding subscore of 0 or 1. The MMS is a composite score of ulcerative colitis disease activity calculated as the sum of three subscores: SF subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal); RB subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed); ES subscore, based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration)
Time Frame: Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the clinical response measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: 50 mg Miri SC Q4W | Maintenance Period: 100 mg Miri SC Q4W | Maintenance Period: 200 mg Miri SC Q4W | Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC | Maintenance Period: 10 mg/kg Miri IV/100 mg Miri SC | Maintenance Period: 300 mg Miri IV/200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
percentage of participants | 0.0 [0.0 to 79.3] | 75.0 [40.9 to 92.9] | 88.9 [56.5 to 98.0] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 39.0]

4. Secondary Outcome: Percentage of Participants Who Are in MMS Clinical Remission Without the Use of Corticosteroids
Description: Corticosteroid-free clinical remission was defined as an SF subscore = 0 or 1, RB subscore = 0, ES ≤ 1 (excluding friability), and have not received corticosteroids for ≥ 12 weeks in the 52-Week Treatment Period. Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the modified mayo score clinical remission without the use of corticosteroids measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maintenance Period: 10 mg/kg Miri IV/ 100 mg Miri SC: Participants (≤40 kg) who were non responders to miri at week 12 in induction received 10 mg SC Q4W for 12 weeks or discontinued after repeat induction, and then received 100 mg miri (>20 to ≤40 kg weight) SC Q4W through week 48 or until loss of response was confirmed.
- Maintenance Period: 300 mg Miri IV/ 200 mg Miri SC: Participants (>40 kg) who were non responders to miri at week 12 in induction received 300 mg SC Q4W for 12 weeks or discontinued after repeat induction, then received 200 mg miri SC Q4W through week 48 or until loss of response was confirmed.
Arm/Group | Maintenance Period: 50 mg Miri SC Q4W | Maintenance Period: 100 mg Miri SC Q4W | Maintenance Period: 200 mg Miri SC Q4W | Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC | Maintenance Period: 10 mg/kg Miri IV/ 100 mg Miri SC | Maintenance Period: 300 mg Miri IV/ 200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
percentage of participants | 0.0 [0.0 to 79.3] | 62.5 [30.6 to 86.3] | 55.6 [26.7 to 81.1] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 39.0]

5. Secondary Outcome: Percentage of Participants in Clinical Remission Based on the Pediatric Ulcerative Colitis Activity Index (PUCAI)
Description: The PUCAI is a clinician-administered, 6-item questionnaire that measures: abdominal pain; RB; stool consistency; number of stools; nocturnal stools; and activity level. For PUCAI score all items are answered as an average over the 'past 2 days'. A total disease activity score is calculated from 0 to 85, with Severe 65-85; Moderate:35-60; Mild:10-30, and None:<10. The clinician will record the participant or caregiver/legal guardian responses for the PUCAI electronically as source data in the tablet device at appropriate visits. PUCAI clinical remission is defined as a PUCAI score of <10 points.
Time Frame: Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the clinical remission based on the PUCAI measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: 50 mg Miri SC Q4W | Maintenance Period: 100 mg Miri SC Q4W | Maintenance Period: 200 mg Miri SC Q4W | Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC | Maintenance Period: 10 mg/kg Miri IV/100 mg Miri SC | Maintenance Period: 300 mg Miri IV/200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
percentage of participants | 0.0 [0.0 to 79.3] | 75.0 [40.9 to 92.9] | 77.8 [45.3 to 93.7] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 39.0]

6. Secondary Outcome: Percentage of Participants in Clinical Response Based on the PUCAI
Description: PUCAI clinical response is defined as a reduction in baseline PUCAI score of ≥20 points.
Time Frame: Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the clinical response based on the PUCAI measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: 50 mg Miri SC Q4W | Maintenance Period: 100 mg Miri SC Q4W | Maintenance Period: 200 mg Miri SC Q4W | Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC | Maintenance Period: 10 mg/kg Miri IV/100 mg Miri SC | Maintenance Period: 300 mg Miri IV/200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
percentage of participants | 0.0 [0.0 to 79.3] | 75.0 [40.9 to 92.9] | 88.9 [56.5 to 98.0] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 39.0]

7. Secondary Outcome: Percentage of Participants in Endoscopic Remission
Description: Endoscopic remission at week 52 is defined as achieving a Mayo endoscopic subscore of 0 or 1 (excluding friability) at Week 52. ES subscore is based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
Time Frame: Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the endoscopic remission measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: 50 mg Miri SC Q4W | Maintenance Period: 100 mg Miri SC Q4W | Maintenance Period: 200 mg Miri SC Q4W | Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC | Maintenance Period: 10 mg/kg Miri IV/100 mg Miri SC | Maintenance Period: 300 mg Miri IV/200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
percentage of participants | 0.0 [0.0 to 79.3] | 62.5 [30.6 to 86.3] | 55.6 [26.7 to 81.1] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 39.0]

8. Secondary Outcome: Percentage of Participants in Symptomatic Remission
Description: Symptomatic remission at week 52 is defined as a Mayo score for RB=0, SF=0 or 1 with ≥ 1 point decrease from baseline.
  SF subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal).
  RB subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed).
Time Frame: Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the symptomatic remission measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: 50 mg Miri SC Q4W | Maintenance Period: 100 mg Miri SC Q4W | Maintenance Period: 200 mg Miri SC Q4W | Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC | Maintenance Period: 10 mg/kg Miri IV/100 mg Miri SC | Maintenance Period: 300 mg Miri IV/200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
percentage of participants | 0.0 [0.0 to 79.3] | 75.0 [40.9 to 92.9] | 66.7 [35.4 to 87.9] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 39.0]

9. Secondary Outcome: Height Velocity (in Centimeters/Year)
Description: Observed height velocity by gender and age group was calculated. Age groups for which this was summarized were 2 to <8, 8 to <12, and 12 to <18. Observed height velocity by gender and age group was calculated at baseline according to the following formula: (Present Height [cm] - Previous Height [cm])/Interval (months) Between Measurements × 12.
Time Frame: Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the height velocity measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Mean (Standard Deviation); unit: centimeter per year (cm/year)
Groups:
- OL Induction and Maintenance Period: 5 mg/kg Miri IV: Participants (≤40 kg weight) received 5 mg/kg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks followed by IV or SC mirikizumab based on their week 12 response status and weight through week 48 or until loss of response was confirmed.
- OL Induction and Maintenance Period: 10 mg/kg Miri IV: Participants (≤40 kg weight) received 10 mg/kg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks followed by IV or SC mirikizumab based on their week 12 response status and weight through week 48 or until loss of response was confirmed.
- OL Induction and Maintenance Period: 300 mg Miri IV: Participants (>40 kg weight) received 300 mg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks followed by IV or SC mirikizumab based on their week 12 response status and weight through week 48 or until loss of response was confirmed.
Arm/Group | OL Induction and Maintenance Period: 5 mg/kg Miri IV | OL Induction and Maintenance Period: 10 mg/kg Miri IV | OL Induction and Maintenance Period: 300 mg Miri IV
Number analyzed (Participants) | 10 | 5 | 11
centimeter per year (cm/year)
  Female: 2 - <8 years: number analyzed (Participants) | 1 | 0 | 0
  Female: 2 - <8 years | NA (NA) — Individual value = 7.85 |  |
  Female: 8 - <12 years: number analyzed (Participants) | 2 | 0 | 0
  Female: 8 - <12 years | 8.65 (3.2) |  |
  Female: 12 - <18 years: number analyzed (Participants) | 3 | 2 | 2
  Female: 12 - <18 years | 4.54 (4.2) | 4.14 (1.3) | 2.97 (0.2)
  Male: 2 - <8 years: number analyzed (Participants) | 1 | 0 | 0
  Male: 2 - <8 years | NA (NA) — Individual value = 7.72 |  |
  Male: 8 - <12 years: number analyzed (Participants) | 0 | 1 | 0
  Male: 8 - <12 years |  | NA (NA) — Individual value = 3.64 |
  Male: 12 - <18 years: number analyzed (Participants) | 2 | 1 | 4
  Male: 12 - <18 years | 12.67 (1.0) | NA (NA) — Individual value = 3.64 | 3.65 (4.3)

10. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from Baseline in body weight by gender and age group was calculated.
Time Frame: Baseline, Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the body weight measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | OL Induction and Maintenance Period: 5 mg/kg Miri IV | OL Induction and Maintenance Period: 10 mg/kg Miri IV | OL Induction and Maintenance Period: 300 mg Miri IV
Number analyzed (Participants) | 10 | 5 | 11
kg
  Female: 2 - <8 years: number analyzed (Participants) | 1 | 0 | 0
  Female: 2 - <8 years | NA (NA) — Individual value = 5.1 |  |
  Female: 8 - <12 years: number analyzed (Participants) | 2 | 0 | 0
  Female: 8 - <12 years | 8 (1.1) |  |
  Female: 12 - <18 years: number analyzed (Participants) | 3 | 2 | 2
  Female: 12 - <18 years | 9 (7.1) | 9 (3.5) | 8 (2.7)
  Male: 2 - <8 years: number analyzed (Participants) | 1 | 0 | 0
  Male: 2 - <8 years | NA (NA) — Individual value = 1.3 |  |
  Male: 8 - <12 years: number analyzed (Participants) | 0 | 1 | 0
  Male: 8 - <12 years |  | NA (NA) — Individual value = 3 |
  Male: 12 - <18 years: number analyzed (Participants) | 2 | 1 | 4
  Male: 12 - <18 years | 13 (11.6) | NA (NA) — Individual value = 3.6 | 2 (3.2)

11. Secondary Outcome: Percentage of Participants With Histologic-Endoscopic Mucosal Remission
Description: Histologic-endoscopic mucosal remission is defined as achieving both histologic remission and endoscopic remission. Histologic remission is defined as Geboes histological subscores of 0 for parameters: 2B (neutrophils in lamina propria), 3 (neutrophils in epithelium), 4 (crypt destruction), and 5 (erosion or ulceration).
Time Frame: Week 52
Population: mITT: All randomized participants who received at least one dose of study drug and who had the histologic-endoscopic mucosal remission measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: 50 mg Miri SC Q4W | Maintenance Period: 100 mg Miri SC Q4W | Maintenance Period: 200 mg Miri SC Q4W | Maintenance Period: 10 mg/kg Miri IV/50 mg Miri SC | Maintenance Period: 10 mg/kg Miri IV/100 mg Miri SC | Maintenance Period: 300 mg Miri IV/200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
percentage of participants | 0.0 [0.0 to 79.3] | 62.5 [30.6 to 86.3] | 44.4 [18.9 to 73.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 39.0]

12. Secondary Outcome: Change From Baseline in 7-day Average of Abdominal Pain Numeric Rating Scale (NRS) Score at Week 12
Description: The Abdominal Pain NRS is a single participant-reported item that measures the "worst abdominal pain in the past 24 hours" using a 6-point scale ranging from 0 (no pain) to 5 (worst possible pain) for 8-11 years old, and 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain) for children < 8 years old as completed by a caregiver and those 12-17 years old. Abdominal Pain NRS Score is calculated by averaging data from all available daily diary entries of abdominal pain NRS for a 7 day period. A negative change from baseline indicates improvement in the participant's Abdominal Pain NRS.
Time Frame: Baseline, Week 12
Population: mITT: All randomized participants who received at least one dose of study drug and who had the 7-day average of Abdominal Pain NRS measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Open Label Induction Period: 5 mg/kg Miri IV: Participants (≤40 kg weight) received 5 mg/kg mirikizumab given as an IV infusion Q4W on weeks 0, 4, 8 for 12 weeks.
Arm/Group | Open Label Induction Period: 5 mg/kg Miri IV | Open Label Induction Period: 10 mg/kg Miri IV | Open Label Induction Period: 300 mg Miri IV
Number analyzed (Participants) | 10 | 5 | 11
score on a scale
  2 - <8 years: number analyzed (Participants) | 3 | 0 | 0
  2 - <8 years | -3 (2.1) |  |
  8 - <12 years: number analyzed (Participants) | 2 | 1 | 0
  8 - <12 years | -3 (2.1) | NA (NA) — Individual value = -2 |
  12- <18 years: number analyzed (Participants) | 5 | 3 | 10
  12- <18 years | -4 (2.7) | -2 (1.5) | -1 (2.8)

13. Secondary Outcome: Change From Baseline in 7-day Average of Abdominal Pain NRS Score at Week 52
Description: as for outcome 12
Time Frame: Baseline, Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OL Maintenance Period: 50 mg Miri SC: Participants (≤20 kg weight) who were responders to mirikizumab at week 12 in induction received 50 mg subcutaneously (SC) Q4W from week 12 through week 48 or until loss of response was confirmed.
Arm/Group | OL Maintenance Period: 50 mg Miri SC | OL Maintenance Period: 100 mg Miri SC | OL Maintenance Period: 200 mg Miri SC | OL Maintenance Period: NR: 10 mg/kg Miri IV/50 mg Miri SC | OL Maintenance Period: NR: 10 mg/kg Miri IV/100 mg Miri SC | OL Maintenance Period: NR: 300 mg Miri IV /200 mg Miri SC
Number analyzed (Participants) | 1 | 8 | 9 | 1 | 1 | 6
score on a scale
  2 - <8 years: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 0
  2 - <8 years | NA (NA) — Individual value = -2 | NA (NA) — Individual value = -6 |  | 0 (0) |  |
  8 - <12 years: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0
  8 - <12 years |  | -2 (1.0) |  |  |  |
  12- <18 years: number analyzed (Participants) | 0 | 3 | 8 | 0 | 1 | 6
  12- <18 years |  | -5 (3.1) | -4 (2.4) |  | NA (NA) — Individual value = -3 | 0 (2.6)

ADVERSE EVENTS:
Time Frame: Induction Period (Up to 12 Weeks), Induction and Maintenance Period (Up to 52 Weeks)
Description: All participants who received at least one dose were analyzed by initial treatment group assignment. Induction, combined induction and maintenance periods were pre-specified for safety analyses; data from the maintenance period alone was not analyzed. Per Stat analysis plan, safety summaries are based on treatment assigned at beginning of induction/maintenance and do not include rescue dosing or weight group changes. Gender specific event denominators were adjusted accordingly.
Groups:
- OL Induction Period: 5 mg/kg Miri IV: Participants (≤40 kg weight) received 5 mg/kg mirikizumab given as an IV infusion every 4 Q4W on weeks 0, 4, 8 for 12 weeks.
Arm/Group | OL Induction Period: 5 mg/kg Miri IV | OL Induction Period: 10 mg/kg Miri IV | OL Induction Period: 300 mg Miri IV | OL Induction and Maintenance Period: 5 mg/kg Miri IV | OL Induction and Maintenance Period: 10 mg/kg Miri IV | OL Induction and Maintenance Period: 300 mg Miri IV
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/11 | 0/10 | 0/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/11 | 0/10 | 2/5 | 1/11
Other Adverse Events (participants affected / at risk) | 8/10 | 2/5 | 8/11 | 9/10 | 5/5 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OL Induction Period: 5 mg/kg Miri IV (N=10) | OL Induction Period: 10 mg/kg Miri IV (N=5) | OL Induction Period: 300 mg Miri IV (N=11) | OL Induction and Maintenance Period: 5 mg/kg Miri IV (N=10) | OL Induction and Maintenance Period: 10 mg/kg Miri IV (N=5) | OL Induction and Maintenance Period: 300 mg Miri IV (N=11)
Appendicitis noninfective (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | OL Induction Period: 5 mg/kg Miri IV (N=10) | OL Induction Period: 10 mg/kg Miri IV (N=5) | OL Induction Period: 300 mg Miri IV (N=11) | OL Induction and Maintenance Period: 5 mg/kg Miri IV (N=10) | OL Induction and Maintenance Period: 10 mg/kg Miri IV (N=5) | OL Induction and Maintenance Period: 300 mg Miri IV (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Growth hormone deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1)
Administration site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (7) | 3 (22)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Puncture site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Immunosuppression (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (7) | 0 (0) | 1 (1) | 3 (8) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/6 (0) | 0/3 (0) | 1/6 (1) | 0/6 (0) | 0/3 (0) | 1/6 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT04004611/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT04004611/SAP_001.pdf